CLINICAL TRIAL: NCT00182949
Title: Genetics and Epidemiology of Aging Associated Conditions in the Sardinian Population (SARDINIA)
Brief Title: Genetics and Epidemiology of Aging Associated Conditions in the Sardinian Population
Status: Completed | Type: Observational
Sponsor: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999904317; 04-AG-N317
Record Dates: First submitted 2005-09-13; First posted 2005-09-16 (Estimated); Last update posted 2018-04-05 (Actual); Status verified 2015-01-02

CONDITIONS: Heart Disease; Physical Frailty; Exaggerated Personality Traits
Keywords: Epidemiology; Genetics; Aging; Sardinian Population; Cardiovascular Diseases; Personality Traits; Frailty
MeSH Terms: conditions — Heart Diseases; Cardiovascular Diseases; Frailty

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Background:

- The island of Sardinia, an Italian region, has a population that is highly interrelated. Researchers have developed the SardiNIA longitudinal study to examine the possible genetic factors that predispose individuals to diseases and to various inherited conditions. In the study, participants will be drawn from four towns in the Ogliastra region (Lanusei, Ilbono, Elini, and Arzana), and their DNA will be analyzed and compared with a long-term assessment of various health-related events. The SardiNIA study is designed to improve understanding of the genetic factors involved in age-associated diseases and disorders, and provide possible points of intervention that may help prevent diseases.

Objectives:

- To conduct a long-term study of genetics and epidemiology in a small and highly interrelated population.

Eligibility:

- Individuals at least 18 years of age (at least 14 years of age for Phase 1 of the study) who live in the province of Ogliastra in eastern Sardinia.

Design:

* This 10-year study will involve three phases: collecting initial blood samples and medical history (years 1 to 4), and two sets of follow-up visits to collect additional data (3 years apart).
* Participants will provide detailed medical history and information for long-term study, primarily involving the following aspects:
* Demographic/family and clinical variables (e.g., medications, fertility, hospitalizations and surgical procedures, age of relatives who are still alive, age and cause of death in deceased relatives) (Phase 1)
* Complete physical examination, including measures of height and weight, blood pressure, and basic heart function (Phase 1)
* Blood and urine samples (Phase 1)
* Heart and lung function tests (Phase 1)
* Assessment of general personality traits and possible history of depression (Phase 1)
* Dietary assessment through a food frequency questionnaire (Phase 1)
* Cognitive tests of attention, memory, and concentration (Phases 1 and 2)
* Frailty-related tests (e.g., hand grip strength, walking speed, bone strength) (Phases 1 and 2)
* Eye examination to test for evidence of disease or macular degeneration (Phases 1 and 2)
* Kidney and thyroid ultrasound (Phases 1, 2, and 3)

DETAILED DESCRIPTION:
The 1,500,000 people of the island of Sardinia arose from a much smaller number, starting thousands of years ago, with very little immigration from outside during that entire period. SardiNIA is a longitudinal study designed under the assumption that in highly interrelated population, such as the Sardinians, discovering the genetic factors that predispose individuals to disease and to other physiological characteristics is easier and more cost-effective. Thus far, group of 6,148 participants from a cluster of 4 towns in the Ogliastra region (Lanusei, Ilbono, Elini, and Arzana) has been assessed for about 100 quantitative traits, including a range of traits related to heart disease, features of personality, frailty, cognition and several blood tests (see Table 1). The DNA from all participants has been analyzed (genotyped) to look for variants of genes that are involved in determining the traits. Up to now, at least one gene has been discovered for each trait, including genes specific for levels of uric acid, fetal hemoglobin, cholesterol, etc. The analyses of genes are continuing, and are being extended to additional traits In addition, to improve the longitudinal perspective of the study, participants will be followed to detect the development on new health-related events or outcomes . This is done in 3 ways: 1) looking at genetic factors determining rates of change of levels of traits like blood pressure with age, based on repeated measures in currently ongoing second visits and planned third visits; 2) seeing which participants do or do not contract particular diseases, to test whether the genes discovered that affect risk factors can help to predict related health problems; and 3) comparing the DNA of disease-free participants in the study to DNA from Sardinian patients affected by particular diseases, to see if the genes already found or additional ones uncovered by the comparisons are involved in those diseases By looking at the development of outcomes, the SardiNIA project (called ProgeNIA for the population) further improves our understanding of the genetic factors involved in age-associated diseases and disorders. Those genes may then provide possible points of intervention that may yield routes to prevention of the diseases.

ELIGIBILITY:
* INCLUSION CRITERIA:

The targeted region for the studies, Ogliastra, is an isolated population of 300,000 in an area enclosed by two mountain ranges and the sea. We will recruit from the 8,500 residents in the towns of Lanusei (the capital of the region), Arzana, Elini and Ilbono, independent of their health status.

EXCLUSION CRITERIA:

At baseline, individuals less than 14 years of age will be excluded from study enrollment. Over the following visits, only individuals 18 and over will be evaluated.

Min Age: 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6926 (Actual)
Dates: Start 2003-11-19; Study Completion 2015-01-02

CONTACTS AND LOCATIONS:
Overall Officials: David A Schlessinger, Ph.D., Principal Investigator — National Institute on Aging (NIA)
Locations (1):
- Italian National Research Council Institute of Neurogenetics and Neuropharmacolo, Lanusei, Italy

REFERENCES:
- [Background] Risch NJ. Searching for genetic determinants in the new millennium. Nature. 2000 Jun 15;405(6788):847-56. doi: 10.1038/35015718. PMID 10866211
- [Background] Liao D, Arnett DK, Tyroler HA, Riley WA, Chambless LE, Szklo M, Heiss G. Arterial stiffness and the development of hypertension. The ARIC study. Hypertension. 1999 Aug;34(2):201-6. doi: 10.1161/01.hyp.34.2.201. PMID 10454441
- [Background] Vaitkevicius PV, Fleg JL, Engel JH, O'Connor FC, Wright JG, Lakatta LE, Yin FC, Lakatta EG. Effects of age and aerobic capacity on arterial stiffness in healthy adults. Circulation. 1993 Oct;88(4 Pt 1):1456-62. doi: 10.1161/01.cir.88.4.1456. PMID 8403292